CLINICAL TRIAL: NCT06173817
Title: The Use of Isocapnic Hyperventilation (iHV) for Treatment of Methanol Poisoned Patients
Acronym: iHV-Met
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulties in working across borders due to sanctions
Sponsor: Oslo University Hospital (Other)
Collaborators: Loghman-Hakim Hospital, Teheran, Iran (Unknown); Shohada-e-Tajrish Hospital, Teheran, Iran (Unknown); Baharloo Hospital, Teheran, Iran (Unknown); Imam Reza Hospital, Mashhad University of Medical Sciences, Iran (Unknown); Khorshid Hospital, Isfahan University of Medical Sciences, Iran (Unknown)
Responsible Party: Principal Investigator, Knut Erik Hovda, MD, PhD, Senior Consultant & Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iHV-Met_2.0; U1111-1277-6360 (Other: WHO UTN); 475313 (Other: Regional Ethics Committee Norway); IRCT20120629010133N5 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2023-11-21; First posted 2023-12-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Methanol Poisoning
Keywords: isocapnic hyperventilation

STUDY DESIGN:
Intervention Model Description: Prospective, single arm study
  * Enrolment target: 30 evaluable patients
  * Intervention: standard of care with sodium bicarbonate and fomepizole, plus iHV device treatment
  * Rescue therapy: haemodialysis at investigators discretion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isocapnic hyperventilation (iHV) (Experimental): Loading dose of fomepizole on clinical suspicion; A) History of intake of alcohol of unknown/illegal origin plus symptoms potentially occurring from methanol, or B) history as above and verified methanol poisonings among people drinking the same alcohol, or C) metabolic acidosis of unknown origin (where methanol cannot be excluded as the cause;or D) a combination of these.
  ● iHV started after a S-methanol concentration > 50 mg/dL is obtained (typically within 4 hours) and initial acidosis is partly or fully corrected by sodium bicarbonate (BD <15mM, HCO3- >10mM)
  Interventions: Device: isocapnic hyperventilation

INTERVENTIONS:
Device: isocapnic hyperventilation — isocapnic hyperventilation (iHV) increases the elimination of methanol to the extent that it could replace haemodialysis for elimination purposes when haemodialysis is not required for the correction of acidosis, and alcohol dehydrogenase (ADH) is completely blocked by an antidote.

SUMMARY:
The projects investigate if treatment with isocapnic hyperventilation can eliminate methanol from the body in a similar manner to dialysis. This is achieved by administering the antidote (fomepizole) and let the patient breathe on a isocapnic hyperventilation device while samples of blood, urine and maybe the breath are collected to measure the contents of methanol and its metabolites.

DETAILED DESCRIPTION:
Isocapnic hyperventilation (iHV) The normal physiology breathing is a careful balance between the number of breaths per minute (rate/min) and the depth of each breath (tidal volume, Vt). Together they make up the minute ventilation (MV), where MV= rate x Vt). To maintain stable homeostasis in the organism, the minute ventilation is closely regulated to maintain adequate uptake of oxygen and adequate elimination of the carbon dioxide (CO2) that is produced by the metabolism. Too low minute ventilation leads to a buildup of CO2 and decrease in blood pH (respiratory acidosis), while hyperventilation (too high minute ventilation) leads to an excess loss of CO2 and increase in blood pH (respiratory alkalosis). The same mechanism will also enable the organism to compensate any metabolic disturbances (up to a certain point): A metabolic acidosis will be counteracted by a hyperventilation, whereas a metabolic alkalosis will be counteracted by a hypoventilation, both with the ultimate goal of keeping the acidity (as given by the pH) as closely regulated as possible.

The concept of isocapnic hyperventilation (iHV) allows the person to hyperventilate while keeping the CO2 within normal limits at the same time. The ClearMate (Thornhill Research Inc., Canada) adds CO2 to the inspired air to compensate to the increased loss induced by the increased minute ventilation. This means that hyperventilation can occur, and a wash-out of volatile substances such as methanol will happen without disrupting the important CO2 balance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, men & women diagnosed with methanol poisoning
* Serum-methanol ≥ 50 mg/dL (16 mM)
* pH ≥ 7.0, and correctable by bicarbonate infusion
* no (newly developed) visual disturbances

Exclusion Criteria:

* Acidosis requiring haemodialysis (pH <7.0), or acidosis that is not responding in spite of aggressive buffer (bicarbonate) treatment within maximum 1-2 hours.
* Comatose patients
* Newly developed visual disturbances
* ADH not fully blocked with antidotes, and not responding to additional dosing of fomepizole. Will be identified by a continuous or increasing anion gap (AG) or Base Excess (BE) on the blood gas machine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-29 (Actual); Primary Completion 2026-01-29 (Actual); Study Completion 2026-01-29 (Actual)

PRIMARY OUTCOMES:
Characterization of methanol elimination kinetics, when iHV is utilized | 0-40 hours
  T1/2 S-methanol (t1-t2) during iHV: Half-life of methanol in blood from start (t1) to end (t2) of treatment with iHV
  T1/2 S-methanol (t0-t1) before iHV): Half-life of methanol in blood from t0 to t1 before start of treatment with iHV for evaluation of individual differences in kinetics

SECONDARY OUTCOMES:
Characterization of methanol elimination kinetics, prior to iHV is utilized | 0-40 hours
  T1/2 S-methanol (t0-t1) before iHV): Half-life of methanol in blood from t0 to t1 before start of treatment with iHV for evaluation of individual differences in kinetics
Serum formate kinetics | 0-40 hours
  T1/2 S-formate before (t0-t1) before and after (t1-t2) (iHV): Half-life of formate in blood from t0 to t1 before start of treatment with iHV for evaluation of individual differences in kinetics
Elimination ratio of methanol | 0-40 hours
  Evaluation of elimination ratio of methanol through breath vs. urine with or without iHV
Elimination ratio of formate | 0-40 hours
  Evaluation of elimination ratio of formate through breath vs. urine with or without iHV
Feasibility of use of iHV in Iran | 0-40 hours
  iHV is new in Iran. The process requires training to be implemented correctly. This will be evaluated by assessing protocol deviations related to iHV equipment and by interviewing study workers on their perceived competency using the iHV equipment.
  This will not be reported in one value, but presented as text and used as an exploratory outcome to guide any future implementation of iHV in Iran
Tolerability by self reporting by patient | 0-40 hours
  Patient tolerability of iHV as self reported by patient
  This will be recorded using a five-level Likert Scale
  1 Did not tolerate iHV at all 2: Tolerated iHV sin shorter periods, but below therapeutic level 3: Barely tolerated iHV enough for therapeutic level 4 Tolerate iHV enough for therapeutic level 5: No discomfort and good toleration of iHV
Implementation of fomepizole in Iran | through study completion, estimated 2 years
  Perception of simplicity of use of fomepizole amongst doctors involved in the study This will be recorded using a five-level Likert Scale
  1 Fomepizole can not be used in the Iranian healthcare system 2: Fomepizole is difficult and require significant extra efforts to be used in the Iranian healthcare system 3: Fomepizole may be used the Iranian healthcare system with some extra effort 4 Fomepizole can easily be used the Iranian healthcare system with little extra effort 5: Fomepizole can easily be used the Iranian healthcare system with no extra effort
Evaluation of fomepizole elimination during iHV | 0-4 hours
  S-fomepizole analyzes from t1-t2. Pending availability of fomepizole analyzes
Length of ICU- and hospital stay | from stdy start to death or discharge ICU, expected average 30 hours
  Length during treatment with iHV
Need for haemodialysis | 0- 40 hours
  Document type and degree of haemodialysis. Indication for such treatment is by the discretion of the local investigator. If S methanol >5mM after 26hrs (T1/2 50-80hrs during fomepizole treatment without haemodialysis (8)) or if patient becomes increasingly acidotic in spite of adequate antidote treatment.
Adverse events | through study completion, estimated 2 years
  Adverse events, including death, will be defined according to Good Clinical Practice guidelines by the International Conference on Harmonization of technical requirements for registration of pharmaceuticals for human use. All adverse events will be registered in this trial and reported in accordance with local regulations in Iran.
  Adverse events also include medical device deficiency of the isocapnic hyperventilation system

CONTACTS AND LOCATIONS:
Overall Officials: Knut Erik Hovda, MD, Ph D, Principal Investigator — The Norwegian CBRNE Centre, Department of Acute Medicine, Oslo University Hospital Oslo, Norway
Locations (1):
- Loghman-Hakim Hospital,, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification will be shared as Investigators discretion.
Supporting Information: Study Protocol, ICF
Time Frame: After publication